CLINICAL TRIAL: NCT05321810
Title: Safety and Effectiveness of Apixaban Compared to Warfarin in Secondary Prevention in Patients With NVAF With a History of Stroke or Transient Ischemic Attack - a Nationwide Retrospective Observational Study Using Claims Data in Japan
Brief Title: Safety and Effectiveness of Apixaban Compared to Warfarin in Secondary Prevention in Patients With Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661176; Secondary prevention (Other: Alias Study Number)
Record Dates: First submitted 2022-04-03; First posted 2022-04-11 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-03

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: Non-valvular atrial fibrillation; Stroke; Apixaban; Warfarin; Secondary prevention
MeSH Terms: conditions — Stroke | interventions — apixaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Warfarin cohort (Reference): Patients with NVAF treated with warfarin
  Interventions: Drug: Warfarin
- Apixaban cohort: Patients with NVAF treated with apixaban
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — This is observational study and the patients in the apixaban cohort include those who are exposed to apixaban in the real world settings.
  Groups: Apixaban cohort
Drug: Warfarin — This is observational study and the patients in the warfarin cohort include those who are exposed to warfarin in the real world settings.
  Groups: Warfarin cohort (Reference)

SUMMARY:
The purpose of this study are 1) to characterize the primary and secondary prevention patients, 2) to calculate incidence rates of stroke/SE or major bleeding in each cohort and 3) to investigate for Japanese secondary prevention patients as Real World Evidence (RWE) on the effectiveness and safety of apixaban compared to warfarin in patients with non-valvular atrial fibrillation (NVAF).

DETAILED DESCRIPTION:
Japanese population has shown to have higher rate of incidence of stroke and stroke mortality is also higher. Patients with a history of ischemic stroke are at high risk of recurrence and require more rigorous management to prevent recurrence. The same is true for patients with non-valvular atrial fibrillation (NVAF) and treatment with anticoagulants reduces the risk of recurrent embolic stroke. However, some patients still suffer from recurrent embolic and/or ischemic stroke even if they are on anticoagulants for secondary prevention. In addition to the recurrent stroke, risk of bleeding is also higher in the patients with a history of stroke because they are often chronically treated with antiplatelet agents to prevent recurrence after cerebral infarction and with an anticoagulant after embolic stroke. Concomitant use of anticoagulant and anti-platelet agents is sometimes necessary if patients with AF experience cerebral infarction and the risk of bleedings largely enhances in these patients. Thus, patients in secondary prevention are at higher risk of both recurrent ischemic stroke and more effective and safer antithrombotic therapy should take this into account.

The purpose of this study are 1) to characterize the primary and secondary prevention patients, 2) to calculate incidence rates of stroke/SE or major bleeding in each cohort and 3) to investigate for Japanese secondary prevention patients as RWE on the effectiveness and safety of apixaban compared to warfarin in patients NVAF.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following selection criteria

1. Patients registered in the Medical Data Vision (MDV) database 2008 though 2021.
2. Patients newly with non-valvular atrial fibrillation
3. Patients who newly receive warfarin or apixaban after diagnosis of NVAF
4. Age 20 years or older on the index date
5. Patients who have a history of stroke or transient ischemic attack (TIA) are inclusion criteria only for secondary prevention cohort, otherwise patients will be concluded in the primary prevention cohort.

Exclusion Criteria:

Patients who meet the following exclusion criteria will be excluded from this study

1. Patients with a diagnosis of valvular AF (standard disease code: 8846941), postoperative AF (8847772), AF associated with mechanical valve malfunction (T82.0), mechanical complication of heart valve prosthesis (T82.0), or rheumatic AF (I05-I09) during the baseline period.
2. Patients with a diagnosis of venous thromboembolism (VTE) during the baseline period
3. Patients who are prescribed any anticoagulants before index date.
4. Patients who are prescribed anticoagulants other than warfarin and apixaban on the index date
5. Patients who are continuously hospitalized due to the first incidence of stroke or other serious diseases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary prevention patients who are newly diagnosed with NVAF and initiate anticoagulation therapy with warfarin or apixaban.
Sampling Method: Probability Sample
Enrollment: 193565 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants diagnosed with non-valvular atrial fibrillation (NVAF) who were newly treated with warfarin or apixaban and were registered in Medical Data Vision (MDV) database during 2008 to 2021 (13 years) were included in this retrospective observational study.
Pre-assignment Details: In this study, inverse probability of treatment weighted (IPTW) method was used in analysis of outcome measures to balance participant's characteristics between warfarin and apixaban cohorts (secondary prevention cohort). To avoid sample size inflation and to ensure appropriate estimation of variances, stabilized IPTW (s-IPTW) was used.
Groups:
- Primary Prevention Cohort: Apixaban: Participants without prior diagnosis of stroke who were newly diagnosed with NVAF and initiated apixaban were included in this study cohort.
- Primary Prevention Cohort: Warfarin: Participants without prior diagnosis of stroke who were newly diagnosed with NVAF and initiated warfarin were included in this study cohort.
- Secondary Prevention Cohort: Apixaban: Participants with prior diagnosis of stroke who were newly diagnosed with NVAF and initiated apixaban were included in this study cohort.
- Secondary Prevention Cohort: Warfarin: Participants with prior diagnosis of stroke who were newly diagnosed with NVAF and initiated warfarin were included in this study cohort.
Period: Overall Study
Arm/Group | Primary Prevention Cohort: Apixaban | Primary Prevention Cohort: Warfarin | Secondary Prevention Cohort: Apixaban | Secondary Prevention Cohort: Warfarin
Started | 57560 | 90636 | 18216 | 27153
Completed | 57560 | 90636 | 18216 | 27153
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all those eligible participants who were newly diagnosed with NVAF and initiated anticoagulation therapy with warfarin or apixaban.
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Prevention Cohort: Apixaban | Primary Prevention Cohort: Warfarin | Secondary Prevention Cohort: Apixaban | Secondary Prevention Cohort: Warfarin | Total
Number analyzed (Participants) | 57560 | 90636 | 18216 | 27153 | 193565
Age, Customized [Count of Participants; unit: Participants]
  Less than or equal to 65 years | 7776 | 15795 | 1380 | 3130 | 28081
  66 years to less than or equal to 75 years | 16219 | 28392 | 4557 | 8104 | 57272
  Greater than 75 years | 33565 | 46449 | 12279 | 15919 | 108212
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22759 | 32232 | 6938 | 9453 | 71382
  Male | 34801 | 58404 | 11278 | 17700 | 122183
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of a Composite of Recurrent Stroke or Systemic Embolism (SE) During the Follow-up Period: Secondary Prevention (Balanced) Cohort
Description: Incidence rate was reported as events per 1,000 participant-years. First occurrence of recurrent stroke or SE events after index date during the follow-up period were considered. Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to stroke or SE". Index date was defined as the next day of the day when participants diagnosed with NVAF initiated warfarin or apixaban. The follow up period was the period until the first observation of the earlier of the following from index date: until discontinuation of index oral anticoagulants (OAC), switch of OAC, lack of records, occurrence of stroke, SE, or hemorrhagic events, or elapsing of 2 years from index date.
Time Frame: During follow up period (Data collected between 2008 to 2021 [approximately 13 years])
Population: Full analysis set included all eligible participants. Analysis was performed using sIPTW method to balance participant characteristics among reporting groups. sIPTW method created balanced virtual groups and hence overall number of participants analyzed is different from numbers in participant flow (not balanced).
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Groups:
- Secondary Prevention Cohort (Balanced): Apixaban: Participants with prior diagnosis of stroke who were newly diagnosed with NVAF and initiated apixaban on the index date and were balanced using sIPTW method.
- Secondary Prevention Cohort (Balanced): Warfarin: Participants with prior diagnosis of stroke who were newly diagnosed with NVAF and initiated warfarin on the index date and were balanced using sIPTW method.
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Events Per 1000 Participant-Years | 41.217 [36.274 to 46.834] | 50.581 [45.658 to 56.034]

2. Primary Outcome: Time Course of Proportion of the Incidence of a Composite of Recurrent Stroke or Systemic Embolism (SE)-Free Participants at 0 Month: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at 0 month was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant recurrent stroke or systemic embolism). Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to stroke or SE".
Time Frame: 0 month
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000]

3. Primary Outcome: Time Course of Proportion of the Incidence of a Composite of Recurrent Stroke or Systemic Embolism (SE)-Free Participants at 6 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at 6 months was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant recurrent stroke or systemic embolism). Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to stroke or SE".
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free | 0.971 [0.966 to 0.976] | 0.967 [0.961 to 0.972]

4. Primary Outcome: Time Course of Proportion of the Incidence of a Composite of Recurrent Stroke or Systemic Embolism (SE)-Free Participants at 12 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at 12 months was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant recurrent stroke or systemic embolism). Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to stroke or SE".
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free | 0.953 [0.946 to 0.960] | 0.948 [0.938 to 0.956]

5. Primary Outcome: Time Course of Proportion of the Incidence of a Composite of Recurrent Stroke or Systemic Embolism (SE)-Free Participants at 18 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at 18 months was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant recurrent stroke or systemic embolism). Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to stroke or SE".
Time Frame: 18 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free | 0.942 [0.933 to 0.951] | 0.932 [0.920 to 0.943]

6. Primary Outcome: Time Course of Proportion of the Incidence of a Composite of Recurrent Stroke or Systemic Embolism (SE)-Free Participants at 24 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at 24 months was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant recurrent stroke or systemic embolism). Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to stroke or SE".
Time Frame: 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free | 0.933 [0.921 to 0.942] | 0.915 [0.900 to 0.928]
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p = 0.016, Log Rank; [Not specified]

7. Primary Outcome: Number of Participants With Risk of a Composite of Recurrent Stroke or SE at 0 Month: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of a composite of recurrent stroke (ischemic and hemorrhagic stroke)/SE at 0 month was reported. Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to stroke or SE".
Time Frame: 0 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants | 7796 | 11601

8. Primary Outcome: Number of Participants With Risk of a Composite of Recurrent Stroke or SE at 6 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of a composite of recurrent stroke (ischemic and hemorrhagic stroke)/SE at 6 months was reported. Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to stroke or SE".
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants | 2061 | 2393

9. Primary Outcome: Number of Participants With Risk of a Composite of Recurrent Stroke or SE at 12 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of a composite of recurrent stroke (ischemic and hemorrhagic stroke)/SE at 12 months was reported. Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to stroke or SE".
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants | 1426 | 1670

10. Primary Outcome: Number of Participants With Risk of a Composite of Recurrent Stroke or SE at 18 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of a composite of recurrent stroke (ischemic and hemorrhagic stroke)/SE at 18 months was reported. Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to stroke or SE".
Time Frame: 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants | 1095 | 1272

11. Primary Outcome: Number of Participants With Risk of a Composite of Recurrent Stroke or SE at 24 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of a composite of recurrent stroke (ischemic and hemorrhagic stroke)/SE at 24 months was reported. Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to stroke or SE".
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants | 845 | 1024
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p = 0.013, t-test, 2 sided; Hazard Ratio (HR) = 0.812, 95% CI 2-sided [0.690 to 0.957]; [Not specified]

12. Primary Outcome: Incidence Rate of Major Bleeding During the Follow-up Period: Secondary Prevention (Balanced) Cohorts
Description: Incidence rate was reported as events per 1,000 participant-years. First occurrence of major bleeding after index date during the follow-up period was considered. Major bleeding, was defined as any bleeding which required hospitalization for treatment (the primary reason for the hospitalization was to treat the bleeding). Index date was defined as the next day of the day when participants diagnosed with NVAF initiated warfarin or apixaban. The follow up period was the period until the first observation of the earlier of the following from index date: until discontinuation of index OAC, switch of OAC, lack of records, occurrence of stroke, SE, or hemorrhagic events, or elapsing of 2 years from index date.
Time Frame: During follow up period (Data collected between 2008 to 2021 [approximately 13 years])
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Events Per 1000 Participant-Years | 28.351 [24.318 to 33.054] | 39.083 [34.793 to 43.903]

13. Primary Outcome: Time Course of Proportion of Incidence of Major Bleeding-Free Participants at 0 Month: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at 0 month was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant major bleeding). Major bleeding, was defined as any bleeding which required hospitalization for treatment (the primary reason for the hospitalization was to treat the bleeding).
Time Frame: 0 month
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000]

14. Primary Outcome: Time Course of Proportion of Incidence of Major Bleeding-Free Participants at 6 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at 6 months was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant major bleeding). Major bleeding, was defined as any bleeding which required hospitalization for treatment (the primary reason for the hospitalization was to treat the bleeding).
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free | 0.983 [0.979 to 0.986] | 0.976 [0.970 to 0.980]

15. Primary Outcome: Time Course of Proportion of Incidence of Major Bleeding-Free Participants at 12 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at 12 months was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant major bleeding). Major bleeding, was defined as any bleeding which required hospitalization for treatment (the primary reason for the hospitalization was to treat the bleeding).
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free | 0.968 [0.961 to 0.974] | 0.963 [0.955 to 0.970]

16. Primary Outcome: Time Course of Proportion of Incidence of Major Bleeding-Free Participants at 18 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at 18 months was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant major bleeding). Major bleeding, was defined as any bleeding which required hospitalization for treatment (the primary reason for the hospitalization was to treat the bleeding).
Time Frame: 18 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free | 0.958 [0.950 to 0.966] | 0.949 [0.938 to 0.958]

17. Primary Outcome: Time Course of Proportion of Incidence of Major Bleeding-Free Participants at 24 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at 24 months was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant major bleeding). Major bleeding, was defined as any bleeding which required hospitalization for treatment (the primary reason for the hospitalization was to treat the bleeding).
Time Frame: 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free | 0.948 [0.937 to 0.957] | 0.932 [0.918 to 0.944]
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p = 0.002, Log Rank; [Not specified]

18. Primary Outcome: Number of Participants With Risk of Major Bleeding at 0 Month: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of major bleeding at 0 month was reported. Major bleeding, was defined as any bleeding which required hospitalization for treatment (the primary reason for the hospitalization was to treat the bleeding).
Time Frame: 0 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants | 7796 | 11601

19. Secondary Outcome: Incidence Rate of Recurrent Cardiogenic Cerebral Embolism During the Follow-up Period: Secondary Prevention (Balanced) Cohorts
Description: Incidence rate was reported as events per 1,000 participant-years. First occurrence of recurrent cardiogenic cerebral embolism after index date during the follow-up period were considered. Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to cardiogenic cerebral embolism". Index date was defined as the next day of the day when participants diagnosed with NVAF initiated warfarin or apixaban. The follow up period was the period until the first observation of the earlier of the following from index date: until discontinuation of index OAC, switch of OAC, lack of records, occurrence of stroke, SE, or hemorrhagic events, or elapsing of 2 years from index date.
Time Frame: During follow up period (Data collected between 2008 to 2021 [approximately 13 years])
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Events Per 1000 Participant-Years | 10.355 [8.043 to 13.332] | 17.893 [15.086 to 21.222]

20. Secondary Outcome: Time Course of Proportion of Incidence of Recurrent Cardiogenic Cerebral Embolism-Free Participants: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at specified time points was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant recurrent cardiogenic cerebral embolism). Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to cardiogenic cerebral embolism ".
Time Frame: 0 month, 6 months, 12 months, 18 months and 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free
  0 Month | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000]
  6 Months | 0.991 [0.987 to 0.993] | 0.989 [0.985 to 0.992]
  12 Months | 0.988 [0.983 to 0.991] | 0.981 [0.974 to 0.986]
  18 Months | 0.984 [0.978 to 0.988] | 0.971 [0.962 to 0.978]
  24 Months | 0.981 [0.975 to 0.986] | 0.967 [0.957 to 0.975]
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p < 0.001, Log Rank; [Not specified]

21. Secondary Outcome: Number of Participants With Risk of Recurrent Cardiogenic Cerebral Embolism: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of recurrent cardiogenic cerebral embolism was reported. Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to cardiogenic cerebral embolism".
Time Frame: 0 month, 6 months, 12 months, 18 months and 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants
  0 Month | 7796 | 11601
  6 Months | 2088 | 2427
  12 Months | 1460 | 1701
  18 Months | 1119 | 1293
  24 Months | 863 | 1047
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p < 0.001, t-test, 2 sided; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.420 to 0.773]; [Not specified]

22. Secondary Outcome: Incidence Rate of Recurrent Cerebral Infarction During the Follow-up Period: Secondary Prevention (Balanced) Cohorts
Description: Incidence rate was reported as events per 1,000 participant-years. First occurrence of recurrent cerebral infarction after index date during the follow-up period were considered. Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to cerebral infarction". Index date was defined as the next day of the day when participants diagnosed with NVAF initiated warfarin or apixaban. The follow up period was the period until the first observation of the earlier of the following from index date: until discontinuation of index OAC, switch of OAC, lack of records, occurrence of stroke, SE, or hemorrhagic events, or elapsing of 2 years from index date.
Time Frame: During Follow up period (Data collected between 2008 to 2021 [approximately 13 years])
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Events Per 1000 Participant-Years | 15.481 [12.581 to 19.048] | 13.430 [11.026 to 16.358]

23. Secondary Outcome: Time Course of Proportion of Incidence of Recurrent Cerebral Infarction-Free Participants: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at specified time points was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant recurrent cerebral infarction). Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to cerebral infarction".
Time Frame: 0 month, 6 months, 12 months, 18 months and 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Groups:
- Primary Prevention Cohort (Balanced): Apixaban: Participants with prior diagnosis of stroke who were newly diagnosed with NVAF and initiated apixaban on the index date and were balanced using sIPTW method.
- Primary Prevention Cohort (Balanced): Warfarin: Participants with prior diagnosis of stroke who were newly diagnosed with NVAF and initiated warfarin on the index date and were balanced using sIPTW method.
Arm/Group | Primary Prevention Cohort (Balanced): Apixaban | Primary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free
  0 Month | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000]
  6 Months | 0.990 [0.987 to 0.992] | 0.989 [0.985 to 0.992]
  12 Months | 0.981 [0.976 to 0.986] | 0.984 [0.978 to 0.988]
  18 Months | 0.976 [0.970 to 0.982] | 0.980 [0.973 to 0.986]
  24 Months | 0.973 [0.965 to 0.979] | 0.977 [0.968 to 0.983]
Statistical Analysis 1: Comparison: Primary Prevention Cohort (Balanced): Apixaban vs Primary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p = 0.350, Log Rank; [Not specified]

24. Secondary Outcome: Number of Participants With Risk of Recurrent Cerebral Infarction: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of recurrent cerebral infarction was reported. Recurrent meant "once participants were discharged from the hospital and became outpatients and then rehospitalized due to cerebral infarction".
Time Frame: 0 month, 6 months, 12 months, 18 months and 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants
  0 Month | 7796 | 11601
  6 Months | 2082 | 2414
  12 Months | 1447 | 1691
  18 Months | 1110 | 1293
  24 Months | 856 | 1046
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p = 0.324, t-test, 2 sided; Hazard Ratio (HR) = 1.155, 95% CI 2-sided [0.867 to 1.540]; [Not specified]

25. Secondary Outcome: Incidence Rate of Intracranial Hemorrhage During the Follow-up Period: Secondary Prevention (Balanced) Cohorts
Description: Incidence rate was reported as events per 1,000 participant-years. First occurrence of intracranial hemorrhage after index date during the follow-up period were considered. Index date was defined as the next day of the day when participants diagnosed with NVAF initiated warfarin or apixaban. The follow up period was the period until the first observation of the earlier of the following from index date: until discontinuation of index OAC, switch of OAC, lack of records, occurrence of stroke, SE, or hemorrhagic events, or elapsing of 2 years from index date.
Time Frame: During follow up period (Data collected between 2008 to 2021 [approximately 13 years])
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Events Per 1000 Participant-Years | 38.214 [33.476 to 43.623] | 44.868 [40.251 to 50.015]

26. Secondary Outcome: Time Course of Proportion of Incidence of Intracranial Hemorrhage-Free Participants: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at specified time points was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant intracranial hemorrhage).
Time Frame: 0 month, 6 months, 12 months, 18 months and 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free
  0 Month | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000]
  6 Months | 0.974 [0.969 to 0.978] | 0.969 [0.963 to 0.973]
  12 Months | 0.959 [0.951 to 0.965] | 0.958 [0.950 to 0.965]
  18 Months | 0.952 [0.943 to 0.959] | 0.951 [0.941 to 0.959]
  24 Months | 0.944 [0.934 to 0.952] | 0.936 [0.924 to 0.947]
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p = 0.111, Log Rank; [Not specified]

27. Secondary Outcome: Number of Participants With Risk of Intracranial Hemorrhage: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of intracranial hemorrhage was reported.
Time Frame: 0 month, 6 months, 12 months, 18 months and 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants
  0 Month | 7796 | 11601
  6 Months | 2069 | 2401
  12 Months | 1434 | 1675
  18 Months | 1106 | 1279
  24 Months | 854 | 1029
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p = 0.100, t-test, 2 sided; Hazard Ratio (HR) = 0.866, 95% CI 2-sided [0.730 to 1.028]; [Not specified]

28. Secondary Outcome: Incidence Rate of Gastrointestinal Bleeding During the Follow-up Period: Secondary Prevention (Balanced) Cohorts
Description: Incidence rate was reported as events per 1,000 participant-years. First occurrence of gastrointestinal bleeding after index date during the follow-up period were considered. Index date was defined as the next day of the day when participants diagnosed with NVAF initiated warfarin or apixaban. The follow up period was the period until the first observation of the earlier of the following from index date: until discontinuation of index OAC, switch of OAC, lack of records, occurrence of stroke, SE, or hemorrhagic events, or elapsing of 2 years from index date.
Time Frame: During follow up period (Data collected between 2008 to 2021 [approximately 13 years])
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Events Per 1000 Participant-Years | 47.634 [42.257 to 53.696] | 47.876 [43.070 to 53.219]

29. Secondary Outcome: Time Course of Proportion of Incidence of Gastrointestinal Bleeding-Free Participants: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at specified time points was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant gastrointestinal bleeding).
Time Frame: 0 month, 6 months, 12 months, 18 months and 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free
  0 Month | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000]
  6 Months | 0.969 [0.964 to 0.974] | 0.968 [0.962 to 0.974]
  12 Months | 0.953 [0.945 to 0.959] | 0.954 [0.945 to 0.962]
  18 Months | 0.931 [0.920 to 0.941] | 0.931 [0.918 to 0.942]
  24 Months | 0.918 [0.905 to 0.929] | 0.915 [0.899 to 0.928]
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p = 0.979, Log Rank; [Not specified]

30. Secondary Outcome: Number of Participants With Risk of Gastrointestinal Bleeding: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of gastrointestinal bleeding was reported.
Time Frame: 0 month, 6 months, 12 months, 18 months and 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants
  0 Month | 7796 | 11601
  6 Months | 2047 | 2381
  12 Months | 1424 | 1664
  18 Months | 1085 | 1257
  24 Months | 828 | 1007
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p = 0.978, t-test, 2 sided; Hazard Ratio (HR) = 1.002, 95% CI 2-sided [0.854 to 1.177]; [Not specified]

31. Secondary Outcome: Incidence Rate of Intraocular Bleeding During the Follow-up Period: Secondary Prevention (Balanced) Cohorts
Description: Incidence rate was reported as events per 1,000 participant-years. First occurrence of intraocular bleeding after index date during the follow-up period were considered. Index date was defined as the next day of the day when participants diagnosed with NVAF initiated warfarin or apixaban. The follow up period was the period until the first observation of the earlier of the following from index date: until discontinuation of index OAC, switch of OAC, lack of records, occurrence of stroke, SE, or hemorrhagic events, or elapsing of 2 years from index date.
Time Frame: During follow up period (Data collected between 2008 to 2021 [approximately 13 years])
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Events Per 1000 Participant-Years | 3.748 [2.463 to 5.704] | 8.627 [6.741 to 11.040]

32. Secondary Outcome: Time Course of Proportion of Incidence of Intraocular Bleeding-Free Participants: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, probability of participants being event-free at specified time points was reported, which was estimated by using a Kaplan-Meier method. (Here, "event" meant intraocular bleeding).
Time Frame: 0 month, 6 months, 12 months, 18 months and 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Probability of being event free
  0 Month | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000]
  6 Months | 0.998 [0.996 to 0.999] | 0.995 [0.992 to 0.997]
  12 Months | 0.995 [0.992 to 0.997] | 0.991 [0.986 to 0.994]
  18 Months | 0.992 [0.987 to 0.995] | 0.987 [0.980 to 0.991]
  24 Months | 0.991 [0.986 to 0.995] | 0.985 [0.977 to 0.990]
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p < 0.001, Log Rank; [Not specified]

33. Secondary Outcome: Number of Participants With Risk of Intraocular Bleeding: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of intraocular bleeding was reported.
Time Frame: 0 month, 6 months, 12 months, 18 months and 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants
  0 Month | 7796 | 11601
  6 Months | 2097 | 2428
  12 Months | 1462 | 1691
  18 Months | 1118 | 1285
  24 Months | 863 | 1040
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p < 0.001, t-test, 2 sided; Hazard Ratio (HR) = 0.428, 95% CI 2-sided [0.263 to 0.697]; [Not specified]

34. Primary Outcome: Number of Participants With Risk of Major Bleeding at 6 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of major bleeding at 6 months was reported. Major bleeding, was defined as any bleeding which required hospitalization for treatment (the primary reason for the hospitalization was to treat the bleeding).
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants | 2081 | 2412

35. Primary Outcome: Number of Participants With Risk of Major Bleeding at 12 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of major bleeding at 12 months was reported. Major bleeding, was defined as any bleeding which required hospitalization for treatment (the primary reason for the hospitalization was to treat the bleeding).
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants | 1448 | 1685

36. Primary Outcome: Number of Participants With Risk of Major Bleeding at 18 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of major bleeding at 18 months was reported. Major bleeding, was defined as any bleeding which required hospitalization for treatment (the primary reason for the hospitalization was to treat the bleeding).
Time Frame: 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants | 1110 | 1283

37. Primary Outcome: Number of Participants With Risk of Major Bleeding at 24 Months: Secondary Prevention (Balanced) Cohorts
Description: In this outcome measure, number of participants with risk of major bleeding at 24 months was reported. Major bleeding, was defined as any bleeding which required hospitalization for treatment (the primary reason for the hospitalization was to treat the bleeding).
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secondary Prevention Cohort (Balanced): Apixaban | Secondary Prevention Cohort (Balanced): Warfarin
Number analyzed (Participants) | 7796 | 11601
Participants | 850 | 1028
Statistical Analysis 1: Comparison: Secondary Prevention Cohort (Balanced): Apixaban vs Secondary Prevention Cohort (Balanced): Warfarin; Statistical analysis has been presented for all time points from 0 to 24 months; Test type: Other; p = 0.001, t-test, 2 sided; Hazard Ratio (HR) = 0.727, 95% CI 2-sided [0.599 to 0.881]; [Not specified]

ADVERSE EVENTS:
Time Frame: Not applicable as safety data were not collected during the study.
Description: This observational retrospective study retrieved data from MDV database and due to the nature of database individual participant data could not be identified. Thus, the minimum criteria (identifiable participant, identifiable reporter, a suspect product, and event) for reporting an adverse event could not be met, hence safety data were not collected and reported.
Groups:
- Secondary Prevention Cohort: Apixaban: Participants with prior diagnosis of stroke who were newly diagnosed with NVAF and initiated apixaban on the index date were included in this study cohort and their data (for the duration of approximately 13 years, i.e. 2008-2021) available in MDV database was retrospectively observed. Index date was defined as the next day of the day when participants diagnosed with NVAF initiated apixaban.
- Secondary Prevention Cohort: Warfarin: Participants with prior diagnosis of stroke who were newly diagnosed with NVAF and initiated warfarin on the index date were included in this study cohort and their data (for the duration of approximately 13 years, i.e. 2008-2021) available in MDV database was retrospectively observed. Index date was defined as the next day of the day when participants diagnosed with NVAF initiated warfarin.
Arm/Group | Secondary Prevention Cohort: Apixaban | Secondary Prevention Cohort: Warfarin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT05321810/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT05321810/SAP_001.pdf